CLINICAL TRIAL: NCT01216605
Title: Oxytocin and Emotion Recognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: X01A-DO1312/1-1; DO1312/1-1 (Other Grant/Funding Number: German Research Foundation (DFG))
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Health
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator)
  Interventions: Drug: Syntocinon 24 IU
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Syntocinon 24 IU
  Arms: Oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The present study was designed to investigate the effects of a single dose of synthetic oxytocin on facial emotion recognition in healthy adult man. Pictures of emotional faces are presented very briefly for a few milliseconds in a backward-masking paradigm in order to vary the level of awareness. In a randomized placebo-controlled between-subject design, recognition performance is compared between a drug (24 IU oxytocin) and a placebo condition. We hypothesize that oxytocin enhances emotion recognition even for facial stimuli processed with limited awareness.

ELIGIBILITY:
Inclusion Criteria:

* Males
* 18 to 40 years of age

Exclusion Criteria:

* Any psychiatric diagnosis life-time
* Somatic disease
* IQ < 85
* Smoker
* Psychoactive medication

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Performance on a facial emotion recognition task | 45 min. following drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Domes, PhD, Principal Investigator — University of Freiburg
Locations (1):
- Department of PSychiatry University of Rostock, Rostock, D, Germany